CLINICAL TRIAL: NCT05832762
Title: Evaluation of Acute Endovascular Treatment in Symptomatic Isolated Cervical Internal Carotid Artery Occlusion
Brief Title: Evaluation of Acute Endovascular Treatment in Symptomatic Isolated Cervical Internal Carotid Artery Occlusion (ETICA)
Acronym: ETICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL21_0527
Record Dates: First submitted 2023-04-14; First posted 2023-04-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic Stroke; Mechanical Thrombectomy; Carotid artery; Stenting; Randomized trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: The protocol is a national, multi-center, prospectively randomized into two parallel (1:1) arms, open to treatment with blinded endpoint trial (PROBE)
Who Masked: Outcomes Assessor
Masking Description: As the therapeutic arm is interventional in the experimental arm, the physicians in charge of the patient and the patients cannot be blinded.
  The mRS score will be evaluated by qualified assessors blinded to the initial treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular treatment + best medical treatment (Experimental): Endovascular treatment associated with the best medical treatment.
  Interventions: Procedure: Endovascular treatment (EVT) + Best medical treatment (BMT)
- best medical treatment (Active Comparator): Best medical treatment alone
  Interventions: Procedure: Best medical treatment (BMT)

INTERVENTIONS:
Procedure: Endovascular treatment (EVT) + Best medical treatment (BMT) — Endovascular treatment (EVT) in the experimental arm can be performed with any recanalization strategy based on the operator's choice, and anatomical and radiological situation: MT using aspiration or stent retriever, with or without stenting (CE-labelled) or angioplasty. In case of acute stenting, the use of antiplatelet drugs will be based on the operator's preference, anatomical situation, and risk of hemorrhage.
  Best medical treatment (BMT) : Administration of drugs is at the treating physician's discretion (for example, intravenous fibrinolysis, anticoagulants, or antiplatelet agents) according to the local standards of care, but not intra-arterial therapies.
  Arms: Endovascular treatment + best medical treatment
Procedure: Best medical treatment (BMT) — Administration of drugs is at the treating physician's discretion (for example, intravenous fibrinolysis, anticoagulants, or antiplatelet agents) according to the local standards of care, but not intra-arterial therapies.
  Arms: best medical treatment

SUMMARY:
Our main hypothesis is that acute EVT associated with best medical treatment is superior to best medical treatment alone, for improving clinical outcomes at 90 days, in patients with mild or severe acute ischemique stroke and diffusion-perfusion or clinical-imaging mismatch, secondary to CICAO.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the superiority of endovascular therapy (EVT) associated with best medical therapy (BMT) (experimental arm) compared to BMT alone (control arm) to increase the functional independence at day 90 3 months (mRS 0-2) in patients with acute cervical isolated internal carotid artery occlusion (CICAO), mild to severe stroke (NIHSS score > 5), and core-perfusion or clinical-imaging mismatch.

Secondary objectives are,(i) to compare the safety of EVT + BMT vs. BMT alone in patients with AIS secondary to CICAO and core-perfusion of clinical imaging mismatch; (ii) to demonstrate the superiority of EVT + BMT vs BMT alone on : the rate of excellent outcome at 3 months (modified Rankin Scale, mRS, score = 0-1),the decrease of the 90-day degree of disability (shift on the mRS combining scores of 5 and 6), the rate of carotid recanalization at 24 hours and at day 90 post-randomization, the cerebral infarct size at 24 hours and at day 90 post-randomization, the early neurological deterioration rate at 24 hours and at day 5- 7 post-randomization, the ischemic recurrences rate at day 90 post-randomization, the early neurological improvement rate at 24h hours post-randomization, the cognitive impairment rate at day 90 post-randomization, the Quality of life at day 90 post-randomization.

One of the secondary objective is also to describe in the experimental group (EVT + BMT), the procedure-related adverse events at day 90 ((Embolism to an intracranial artery, vascular perforation, arterial dissection, access site complication requiring surgical repair or blood transfusion, peri-procedural mortality, device failure).

ELIGIBILITY:
Inclusion Criteria:

* ≥18-year-old patients (no upper age limit)
* Clinical signs consistent with AIS (Acute ischemic stroke)
* NIHSS score >5 at randomization time with time from last seen well to randomization ≤23h, or fluctuating neurological symptoms, defined as recurrent transient attacks and/or progression of neurological deficit within the last 7 days.
* Ischemic stroke confirmed by cerebral imaging (CT: Computed Tomography or MRI:Magnetic Resonance Imaging) or normal imaging with suspected ischemic stroke
* Existence of a mismatch: If perfusion data are available (PWI/CTP), existence of a core-perfusion mismatch, suggestive of carotid hemodynamic mechanism, according to the DEFUSE-3 criteria: mismatch volume ≥15 mL, core volume ≤70 mL, and mismatch ratio ≥1.8 ; if perfusion data are not available, or non interpretable, existence of a clinical-imaging mismatch, defined by an ASPECTS >5 (Alberta Stroke Program Early CT score)
* CICAO (Cervical isolated Internal Carotid Artery Occlusion) all causes (for example dissection, atheroma or undetermined cause) on CTA (Computed Tomography Angiography) or MRA with gadolinium, without associated visible ipsilateral large intracranial occlusion (T or L, M1, M2, A1, A2, P1, P2), <1 h before randomization
* Anticipated possibility to start the EVT procedure (arterial access) within 60 minutes after randomization
* Pre-stroke mRS score ≤2
* Patient or patient's representative has received information about the study and has signed and dated the appropriate Informed Consent or met the criteria for emergency consent, signed by the investigator

Exclusion Criteria:

* CICAO after recent (<1 month) endarterectomy
* Patient with severe or fatal co-morbidities or life expectancy <6 months that will likely interfere with improvement or follow-up or that will render the procedure unlikely to benefit the patient
* Patient unable to come or unavailable for follow-up
* Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations
* Seizures at stroke onset if they make the diagnosis of stroke doubtful and preclude obtaining an accurate baseline NIHSS assessment
* Suspected cerebral vascular disease (e.g., vasculitis) based on the medical history and CTA/MRA
* Pregnancy in progress or planned during the study period, woman who is known to be pregnant or lactating at admission time
* Adult protected by law or patient under guardianship or curators
* Current participation in another investigational drug or device study
* Not affiliated to the French social security system or not beneficiary of such system
* Known contrast or endovascular product life-threatening allergy
* Associated stenosis (≥50%) of the middle cerebral artery ipsilateral to the CICAO
* Chronic CICAO, defined as a known carotid occlusion (on a previous imaging exam) ≥30 days before randomization or high suspicion of chronic CICAO based on medical history and CT/MRI
* Tandem occlusion, defined by cervical ICA occlusion associated with intracranial large vessel occlusion (T- or L-shaped, M1 or M2 portions of the middle cerebral artery, A1 or A2 portions of the anterior cerebral artery, P1 or P2 portions of the posterior cerebral artery)
* Associated ipsilateral large intracranial arterial occlusion
* Prior stenting of the target ICA
* Intracranial stent implanted in the same vascular territory as the CICAO
* Sub-occlusive cervical ICA stenosis on CTA or MRA
* Suspicion of ICA occlusion starting at the petrous, cavernous or intracranial segment with normal cervical portion on non-invasive imaging (MRA or/and CTA)
* Known absence of vascular access
* Suspicion of aortic dissection based on medical history, clinical evaluation or/and imaging
* Sub-occlusive cervical ICA stenosis on CTA or MRA
* Common carotid artery occlusion without ICA occlusion on non-invasive imaging (MRA or/and CTA)
* Evidence of intracranial hemorrhage on CT/MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with favorable functional outcome, defined by a mRS score ≤2 | Day 90 (± 15 days) post-randomization
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.The scale runs from "0" to "6", running from perfect health without symptoms to death.
  The mRS score will be evaluated by qualified assessors blinded to the initial treatment.The blinded evaluator must be familiar with mRS scoring (dedicated training and certification). If a participant is unable to attend in-person the follow-up visit at day 90 (±15), mRS scoring can be done by telephone by a qualified investigator.

SECONDARY OUTCOMES:
The degree of disability at day 90 (±15) post-randomization (shift on the mRS combining scores of 5 and 6) | Day 90 (± 15 days) post-randomization
  The mRS score will be evaluated by qualified assessors blinded to the initial treatment.The blinded evaluator must be familiar with mRS scoring (dedicated training and certification). If a participant is unable to attend in-person the follow-up visit at day 90 (±15), mRS scoring can be done by telephone by a qualified investigator.
Change in NIHSS score at 24 (-6/+12) hours post-randomization. | 24h (-6/+12) post-randomization
  NIHSS score is "the National Institutes of Health Stroke Scale". The NIHSS is composed of 11 items, each of which scores a specific ability between 0 and 4. For each item, a score of 0 typically indicates normal function, while higher scores are indicative of some level of impairment. The individual scores for each item are summed to calculate the patient's total NIHSS score. The maximum possible score is 42, and the minimum score is 0.
Quality of life at day 90 (±15) post-randomization assessed with the EuroQol 5D-5L | Day 90 (± 15 days) post-randomization
  Assessed with the EuroQol 5D-5L which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Cognitive function at day 90 (±15) post-randomization, evaluated with the Montreal Cognitive assessment (MoCA test). | Day 90 (±15 days) post randomization
  The MoCA test is the Montreal Cognitive Assessment measuring the neurocognitive function. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal. This test covers orientation, short-term memory, focus and spatial awareness, language, concentration and clock drawing test.
Carotid artery revascularization rate | randomization
  Assessed by angiography in the experimental arm, defined by complete recanalization or residual carotid artery stenosis <50%
Carotid artery recanalization rate | 24 (-6/+12) hours post randomization
  Assessed by MRA with gadolinium or CTA, defined as complete recanalization or residual carotid artery stenosis <50%
Carotid artery recanalization rate | Day 90 (± 15 days) post-randomization
  Assessed by MRA with gadolinium or CTA, defined as complete recanalization or residual carotid artery stenosis <50%
Infarct volume | 24 (-6/+12) hours post randomization
  Measured by magnetic resonance angiography (MRI, FLAIR) or computed tomography (CT).
Infarct volume | Day 90 (± 15 days) post randomization
  Measured by magnetic resonance angiography (MRI, FLAIR) or computed tomography (CT).
Early neurological improvement | Day 0 - 24 hours post randomization
  Early neurological improvementis defined by an NIHSS score of 0-2 at 24 hours or a ≥8-point decrease of the NIHSS score at 24 hours compared with baseline.
Incidence of all-cause mortality at day 90 | Day 90 (± 15 days) post randomization
  Incidence of all-cause mortality at day 90
Rate of symptomatic intracranial hemorrhage | 24 (-6/+12) hours post-randomization
  According to the Heidelberg Bleeding classification by cerebral imaging
Incidence of procedure/device-related adverse events | Day 30 (±5 days) post randomization
  In the experimental group (EVT + BMT)
Early neurological deterioration rate | 24 hours post-randomization
  NIHSS score increase by ≥4 points
Neurological deterioration rate | Day 5-7 post randomization
  NIHSS score increase by ≥4 points
Rapid NIHSS worsening | Admission - day 5/day 7/discharge (if earlier)
  NIHSS score increase by ≥10 points
Degree of disability at day 30 post-randomization (shift on the mRS combining scores of 5 and 6) | Day 30 (±5 days) post randomization
  The mRS score will be evaluated by qualified assessors.The evaluator must be familiar with mRS scoring (dedicated training and certification). If a participant is unable to attend in-person the follow-up visit at day 30, mRS scoring can be done by telephone by a qualified investigator.
Incidence of symptomatic intracranial hemorrhage according to the SITS-MOST | Day 90 (±15 days) post randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology/ Stroke Unit, Hôpital Gui de Chauliac, Montpellier, Fance, France